CLINICAL TRIAL: NCT01439789
Title: A Phase III, Multi-center,Randomized, Double-blind, Based on Standard Therapy, Placebo-controlled Study of the Efficacy/Safety of Recombinant Human Neuregulin-1β in Patients With Chronic Systolic Heart Failure
Brief Title: Study of Efficacy on NT-proBNP of Recombinant Human Neuregulin-1 in Chronic Heart Failure Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor has designed another study with different endpoint to replace the current study
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-01-304
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2012-07

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; rhNRG-1; NT-proBNP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhNRG-1 (Active Comparator): Recombinant human neuregulin-1 administration in addition to basic therapy of chronic heart failure
  Interventions: Drug: rhNRG-1
- Plaebo (Placebo Comparator): Excipient placebo in addition to basic therapy of chronic heart failure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhNRG-1 — day1~day10:0.6ug/kg/day,10hours per day for vein infusion
  Arms: rhNRG-1
Drug: Placebo — day1~day10:0.6ug/kg/day,10hours per day for vein infusion
  Arms: Plaebo

SUMMARY:
Multi-center, randomized, double-blind , placebo parallel controlled, standard therapy based phase III clinical trial, to evaluate the efficacy of recombinant human neuregulin-1 on serum NT-proBNP, as well as safety in patients with chronic heart failure.

DETAILED DESCRIPTION:
N-terminal proNBP (NT-proBNP) has been proved to be an independent prognostic factor for the long-term prognosis of chronic heart failure patients.RhNRG-1(recombinant human neuregulin-1)directly works on the cardiomyocytes and restored the normal structure and function of it. It has been found that rhNRG-1 effectively decreased the serum level of NT-proBNP,and is tolerated in the effective dosages groups.The aim of this phase III trial is to further confirm in large population that rhRNG-1 administration can effectively decrease the serum level of NT-proBNP and is tolerated in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75, both sex.
2. Left ventricular ejection fraction (LVEF)≤40% (ECHO).
3. NYNA functional class II~III.
4. Definitely diagnosed with chronic systolic heart failure (including medical records, symptoms and physical signs)and clinical symptom is steadily in the latest 1 month.
5. Receiving standard basic treatment of heart failure, has reached the objective dosage or the highest tolerated dosage for at least 1 month, or the dosage has not been changed for at least 1 month.
6. Capable of signing the informed consent form.

Exclusion Criteria:

1. Patients with acute myocardial infarction, Hypertrophic cardiomyopathy, constrictive pericarditis, significant valvular pathological change or congenital heart diseases, severe pulmonary artery hypertension.
2. Ischemic heart failure without recanalization or with recanalization in recent six months.
3. Cardiac surgery or cerebrovascular accident within recent six months.
4. Preparing for heart transplantation or has received CRT treatment.
5. Serious hepatic or renal dysfunction caused by organic pathological changes (Cr>2.0mg/dl, AST or ALT 5 times above the normal upper limit).
6. Patients need mechanical ventilation.
7. Systolic blood pressure <90mmHg or >160mmHg.
8. Patients with acute hemodynamic disorder or decompensation in the last 1 month.
9. Serious ventricular arrhythmia (multi-morphological premature ventricular contraction, frequent paroxysmal ventricular tachycardia).
10. Serum potassium <3.2 mmol/L or >5.5 mmol/L.
11. Pregnant or plan to pregnant.
12. Unmarried or married but not procreated women at child-bearing age.
13. Subject with a life expectancy less than 6 months as assessed by the investigator.
14. Patients who participated in any clinical trial in the recent three months.
15. History of any malignancy or suffering from cancer,or biopsy proven pre-malignant condition (eg DICS or cervical atypia).
16. Evidence (physical examination,CXR,ECHO or other tests) shows some active malignancy or adenoidal hypertrophy or neoplasm has effect on heart function or endocrine system, eg pheochromocytoma or hyperthyroidism.
17. Judging by the investigator, the patients could not complete the study or adhere to the study requirements (due to the management reasons or others).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
NT-proBNP | 30 days

SECONDARY OUTCOMES:
NT-proBNP | 90 days
Six Minutes Walk Distance | 30 days and 90 days
NYHA classification | 30 days and 90 days
Quality of Life | 30 days and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, MD, Ph.D, Principal Investigator — Cardiovascular Institute and Fuwai Hospital
Locations (21):
- China (21):
  - Cardiovascular Institute and Fuwai Hospital, Beijing, Beijing Municipality
  - Bethune Peace Hospital, Shijiazhuang, Hebei
  - Teda International Cardiovascular Hospital, Tianjin, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Sichuan Provincial People's Hospital, Chengdu, Jiangsu
  - The Second Hospital affiliated to Suzhou University, Suzhou, Jiangsu
  - North Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Affiliate Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Hospital affiliated to Dalian Medical University, Dalian, Liaoning
  - The first affiliated hospital of Liaoning medical college, Jinzhou, Liaoning
  - Liaoning Provincial People's Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - The Xinqiao Hospital of Third Military Medical University, Chongqing, Sichuan
  - Kunming General Hospital of Chengdu Military Region, Kunming, Yunnan